CLINICAL TRIAL: NCT05176691
Title: A Multicenter, Open-label, Phase 1 Study Evaluating the Safety and Tolerability of HMPL-760 in Patients With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) or Other Non-Hodgkin Lymphoma (NHL)
Brief Title: HMPL-760 Safety and Tolerability Study in Patients With Previously Treated CLL/SLL or NHL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: HUTCHMED has decided to discontinue the HMPL 760 study.
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-760-GLOB1
Record Dates: First submitted 2021-11-19; First posted 2022-01-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: CLL/SLL; NHL; MCL; MZL; Lymphoplasmacytic Lymphoma; Waldenstrom Macroglobulinemia; Follicular Lymphoma; DLBCL; Richter Syndrome
Keywords: Lymphoplasmacytic lymphoma/Waldenstrom's macroglobulinemia; Chronic lymphocytic leukemia; Non-Hodgkin lymphoma; Mantle cell lymphoma; Marginal zone lymphoma; Follicular lymphoma; Diffuse large B-cell lymphoma; BTK inhibitor
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients to receive HMPL-760 daily.
  Interventions: Drug: HMPL-760

INTERVENTIONS:
Drug: HMPL-760 — Administered orally QD for 28-day cycles

SUMMARY:
An open label single-arm clinical trial to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of HMPL-760 in patients with previously treated CLL/SLL or NHL

DETAILED DESCRIPTION:
HMPL-760 is a highly potent, selective, and reversible inhibitor against BTK, which would be studied in B-cell malignancy carrying either BTK(WT) or BTK(C481S).

This is a phase 1, open-label, multicenter, single-arm study to evaluate safety, tolerability, PK, PD, and preliminary efficacy of HMPL-760 in patients with previously treated CLL/SLL or NHL

The study consists of 2 parts:

Part 1- Dose Escalation to determine MTD and/or RP2D of HMPL-760

Part 2- Dose Expansion to characterize the safety and tolerability of HMPL-760

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1;
* Histologically confirmed NHL or CLL with disease progression or intolerance to either ≥2 prior regimens. Patients with CLL/SLL and indolent NHL must meet criteria for systemic therapy. Patients with gastric extranodal MZL who are H. pylori positive must have failed H. pylori eradication therapy.
* Availability of tumor sample: This may be an archival tissue sample obtained after most recent therapy or a fresh biopsy; if tumor sample is not available for patients in dose escalation, the Sponsor may waive the requirement after discussion.
* Dose expansion stage only: Patients must have been treated with 1 prior regimen containing a BTK inhibitor in cohorts 1 to 5;
* Expected survival of more than 24 weeks as determined by the Investigator.

Exclusion Criteria:

* Patients with primary central nervous system lymphoma.
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) <0.75×109/L
  * Hemoglobin <8 mg/L
  * Platelets <50×109/L
  * Note: In the dose expansion stage, patients with cell counts below the thresholds listed above may be considered eligible if there is documented bone marrow infiltration and Sponsor approval
* Inadequate organ function
* International normalized ratio (INR) >1.5×ULN, activated partial thromboplastin time (aPTT) >1.5×ULN

  - Patients requiring anticoagulation therapy (except vitamin K antagonists [ie, warfarin]) but with a stable INR within the recommended range according to the local guideline are eligible.
* Patients with presence of second primary malignant tumors within the last 2 years, with the exception of the following:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
* Clinically significant history of liver disease, including cirrhosis or current known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV).
* Cancer therapy, including chemotherapy, hormonal therapy, biologic therapy, vaccine, or radiotherapy within 3 weeks prior to initiation of study treatment. For oral targeted therapies, a washout period of 5 half-lives of the agent (minimum 3 days) prior to the initiation of study treatment can be used.
* Any granulocyte colony-stimulating factor treatment/blood transfusion within 7 days before the screening hematology test.
* Prior use of any drug that is a strong inducer or inhibitor of CYP3A4 within 2 weeks prior to initiation of study treatment.
* Prior use of proton pump inhibitors (PPIs) within 5 days of study treatment
* Any transplant within 100 days prior to initiation of study treatment
* Clinically significant active infection or with an unexplained fever.
* Treatment within a clinical study of an investigational agent or using an investigational device within 3 weeks prior to initiation of the current study treatment.
* AEs from prior antineoplastic therapy that have not resolved to grade <1
* Pregnant (positive urine or serum beta human chorionic gonadotropin test) or lactating women.
* New Your Heart Association (NYHA) class II or greater congestive heart failure.

NOTE: Only key inclusion/exclusion criteria are listed. Full details are in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs | Up to 28 days after first dose of study drug
  Adverse event (AE) that meets protocol defined DLT criteria during dose escalation
Incidence of AEs/SAEs | From 1st dose to within 30 days of last dose
  Any untoward medical occurrence associated with the use of study drug
MTD | From 1st dose to within 30 days of last dose
  To evaluate maximum tolerated dose of HMPL-760 in subjects, if reached
RP2D | From 1st dose to within 30 days of last dose
  To determine recommended phase 2 dose of HMPL-760 in subjects

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From 1st dose of study drug to the time of progressive disease, assessed up to 36 months
  ORR is defined as the proportion of subjects achieving partial response and better response during the study
Duration of Response (DoR) | From first dose of study drug to the time of progressive disease, assessed up to 36 months
  DoR is defined as the time between the initial response to therapy and subsequent disease progression or relapse.
Clinical Benefit Rate (CBR) | From 1st dose of study drug to the time of progressive disease, assessed up to 36 months
  CBR is defined as the proportion of subjects achieving objective response or stable disease
Progression-free Survival (PFS) | From 1st dose of study drug to the time of progressive disease, assessed up to 36 months
  PFS is defined as survival without progression of the disease
Maximum Plasma Concentration [Cmax] | From 1st dose to within 30 days of last dose
  To determine the maximum observed plasma concentration of HMPL-760
Chemokines | From 1st dose to within 30 days of last dose
  To observe blood plasma concentrations of chemokines such as CCL22 and CCL3
Phospho-BTK | From 1st dose to within 30 days of last dose
  To observe the whole blood concentrations of phospho-BTK

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Jayaprakash, MBBS, PHD, Study Director — Hutchison Medipharma Limited
Locations (36):
- United States (12):
  - Innovative Clinical Research, Anaheim, California
  - Emory University Hospital, Atlanta, Georgia
  - Tulane Cancer Center, New Orleans, Louisiana
  - Johns Hopkins Clinical Research Center, Baltimore, Maryland
  - AMR Kansas City, Formerly Center for Pharmaceutical Research, an AMR company, Kansas City, Missouri
  - Center For Advanced Medicine, St Louis, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - New York University Langone Med Center. Lab, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - Renovatio Clinical, El Paso, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- France (5):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - Hôpital Saint-Antoine, Paris, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - CHU Poitiers - Hôpital la Milétrie, Poitiers, Vienne
- Israel (4):
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Lazio, Roma
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
- Poland (4):
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Centrum Medyczne Pratia Poznan, Skórzewo
  - MICS Centrum Medyczne Torun, Torun
- Spain (6):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital del Mar, Barcelona
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid